CLINICAL TRIAL: NCT01802723
Title: A Dose Ranging Study of the Safety and Efficacy of LIPO-202 Healthy Patients With Subcutaneous Fat in the Periumbilical Area
Brief Title: Dose Ranging Study
Acronym: RESET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIPO-202-CL-16
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Periumbilical Subcutaneous Adipose Tissue Reduction
MeSH Terms: interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LIPO-202, Low (Experimental): Drug: salmeterol xinafoate
  Interventions: Drug: Drug: salmeterol xinafoate
- LIPO-202, Mid (Experimental): Drug: salmeterol xinafoate
  Interventions: Drug: Drug: salmeterol xinafoate
- LIPO-202, High (Experimental): Drug: salmeterol xinafoate
  Interventions: Drug: Drug: salmeterol xinafoate
- LIPO-202, Placebo (Experimental): Drug: Placebo
  Interventions: Drug: Drug: Placebo

INTERVENTIONS:
Drug: Drug: salmeterol xinafoate
  Other Names: LIPO-202; Salmeterol
  Arms: LIPO-202, High; LIPO-202, Low; LIPO-202, Mid
Drug: Drug: Placebo
  Other Names: Placebo
  Arms: LIPO-202, Placebo

SUMMARY:
Dose Ranging Study

ELIGIBILITY:
Inclusion Criteria:

>18 years of age inclusive Subcutaneous fat in the periumbilical area BMI <30 kg/msq Stable diet and exercise and body weight

Exclusion Criteria:

Prior treatment of subcutaneous fat in the periumbilical area (liposuction, abdominoplasty, etc.) Known hypersensitivity to drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety | 8 weeks treatment
  physical exam, vital signs, clinical assessment of injection, clinical laboratory tests, and adverse events
Change in global clinician abdominal perception scale score (baseline and 9 weeks) | 9 weeks
Change in global patient abdominal perception scale score (baseline and 9 weeks) | 9 weeks
Change in abdominal circumference (baseline and 9 weeks) | 9 weeks
  abdominal circumference

SECONDARY OUTCOMES:
Change in Photonumeric abdominal perception scale score (baseline and 9 weeks) | 9 weeks
Change in Patient Reported Outcome for abdominal perception score (baseline and 9 weeks) | 9 weeks

OTHER OUTCOMES:
Change in subcutaneous abdominal adipose tissue thickness (baseline and 9 weeks) | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murray C Maytom, MBChB, MBA, Study Director — Neothetics, Inc
Locations (22):
- United States (22):
  - United States, California, Beverly Hills, California
  - United States, California, Encinitas, California
  - United States, California, Los Angeles, California
  - United States, California, San Diego, California
  - United States, California, Santa Ana, California
  - United States, Florida, Aventura, Florida
  - United States, Florida, Clearwater, Florida
  - United States, Florida, Lake Worth, Florida
  - United States, Florida, Miami, Florida
  - United States, Florida, Tampa, Florida
  - United States, Illinois, Buffalo Grove, Illinois
  - United States, Illinois, Chicago, Illinois
  - United States, New York, New York, New York
  - United States, New York, Smithtown, New York
  - United States, North Carolina, Chapel Hill, North Carolina
  - United States, North Carolina, Raleigh, North Carolina
  - United States, Tennessee, Nashville, Tennessee
  - United States, Texas, Austin, Texas
  - United States, Texas, Dallas, Texas
  - United States, Texas, Fort Worth, Texas
  - United States, Texas, Houston, Texas
  - United States, Texas, Plano, Texas